CLINICAL TRIAL: NCT05767008
Title: Demonstrate the Water Resistance Properties of Metal Oxide Filters
Brief Title: Water Immersion Studies of a Long-wear Sunscreen to Improve Protection Against Ultraviolet Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanometics (d.b.a. PHD Biosciences) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 43-692
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Sunburn
MeSH Terms: conditions — Sunburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Static and water immersion SPF evaluation (Experimental)
  Interventions: Other: Sunscreen -R43

INTERVENTIONS:
Other: Sunscreen -R43 — Long wear metal oxide particles

SUMMARY:
This study is designed to determine the Sun Protection Factor (SPF) of a test product following 80 Minute Water Immersion methodology defined in Final Monograph - Code of Federal Regulations Title 21 - "Labeling and Effectiveness Testing; Sunscreen Drug Products; Required Labeling Based on Effectiveness Testing", Final Rule, 21 CFR 201.327.(j)

DETAILED DESCRIPTION:
All studies will be carried out in a blind fashion according to FDA guidelines, which describes the number of subjects required to satisfy FDA guidelines and labeling requirements of sunscreens. Human subject selection: Healthy volunteers (n=25) free from systemic or dermatological disorders of Fitzpatrick skin type I, II or III (12 male and 13 female; ages 18 through 55) will be recruited. Rectangular test sites of (30 cm2) on the infrascapular area of the back will be delineated, and inspected to ensure uniform pigmentation, skin tone and texture, and absence of warts, moles, nevi, scars, blemishes and active dermal lesions. SPF determination: A 150 W Xenon Arc Solar Simulator, which produces a continuous UV spectra substantially equivalent to that of natural sunlight will be used and UVB radiation monitored continuously. Measurements will be recorded within 8 mm from the surface of the skin, and the size of the exposure site will be ≥ 0.5 cm2. The Sunscreen or a positive control (8% homosalate) will be applied to subjects evenly in the delineated areas at 2 mg/cm2. Following static exposures, test sample and water resistant controls will be applied on adjacent sites for testing. An unprotected site will receive a series of five UV exposures based upon the previously determined Minimal Erythemal Dose (MED). The UV exposures for each formulation, will be calculated from previously determined MED and the intended SPF. Immersion procedure: Immersion will be conducted in a whirlpool tub with room temperature water circulating at 3450 r.p.m. Following pre-immersion SPF measurements, volunteers will be subjected to 80 min of whirlpool immersion, with SPF measurements taken after air drying at 20, 40, and 80, min. c. Data Analysis and Interpretation: The 80 min time point is chosen as a benchmark for success because the FDA only permits finished sunscreen products to be labeled as water resistant for up to 80 min. All subjects will return to the laboratory sixteen to twenty-four hours post-exposure for a blinded determination of erythema responses, the mean SPF, standard deviation (s) value, and standard error (SE). No attempts to determine the influence of sex or age on the interpretation of results will be undertaken because of Phase I SBIR budgetary and time limitations, and because this is not a requirement of FDA or customers / distribution partners who will purchase the product. The standard deviation (s) will be determined and the upper 5% point was obtained from the t distribution table with n-1 degrees of freedom (t).

ELIGIBILITY:
Inclusion Criteria:

1. Males (n=12) and females (n=13) 18 through 55 years.
2. Fitzpatrick skin type I, II or III.
3. Free from dermatological disorders.

Exclusion Criteria:

1. Volunteers younger than 18 years, or older than 55 years.
2. Volunteers of Fitzpatrick skin type IV or greater.
3. Volunteers with dermatological disorders or the presence of non-uniform pigmentation, skin tone and texture, warts, moles, nevi, scars, blemishes and active dermal lesions at the desired test sites.
4. Volunteers being treated with photosensitizing agents, or have been treated with photosensitizing agents in the prior 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
SPF determination | 80 minutes
  SPF determination before and after water immersion

CONTACTS AND LOCATIONS:
Locations (1):
- Nanometics, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No